CLINICAL TRIAL: NCT04228003
Title: The Effect of Pendulum Glucose Control on GI Symptoms and Glycemic Control in Subjects With Type 2 Diabetes
Brief Title: Pendulum D2D Glucose Control for Adults With Type 2 Diabetes
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: The funding and project never started
Sponsor: University of Southern California (Other)
Collaborators: Pendulum Therapeutics (Industry)
Responsible Party: Principal Investigator, Anne Peters, Professor of Medicine, Clinical Scholar, University of Southern California
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pendulum D2D
Record Dates: First submitted 2020-01-10; First posted 2020-01-14 (Actual); Last update posted 2021-10-07 (Actual); Status verified 2021-09

CONDITIONS: Type2 Diabetes; Gastrointestinal Symptoms

STUDY DESIGN:
Intervention Model Description: The study is a single site, prospective, open label, observational, single arm trial in 30 patients with type 2 diabetes with gastrointestinal complaints.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Pendulum (Experimental): Pendulum Glucose Control formulation for T2D will be taken twice daily - 1 capsule with the morning meal and 1 capsule with the evening meal for 8 weeks with an option of continuing up to 6 months.
  Interventions: Dietary Supplement: Pendulum Glucose Control formulation for T2D

INTERVENTIONS:
Dietary Supplement: Pendulum Glucose Control formulation for T2D — All bacteria contained in the study product formulation are commensal organisms that have been repeatedly documented to inhabit the human GI tract under normal circumstances. Pendulum's Glucose Control Formulation consists of five human commensal microbial strains including butyrate producing and mucin-degrading strains. The organisms were grown under controlled conditions consistent with Good Manufacturing Practices (GMP) and employ no animal-derived products. All ingredients utilized during manufacturing were food grade and qualified as generally recognized as safe (GRAS).
  The product is provided as acid-resistant capsules in bottles that are to be stored refrigerated at 4℃.

SUMMARY:
The study is a single site, prospective, open label, observational, single arm trial in 30 patients with type 2 diabetes with GI complaints using 1 or more oral or injectable anti-hyperglycemic agents to investigate if altering the microbiome though Pendulum T2D dietary supplementation can further enhance the efficacy of the current treatment while reducing the GI associated symptoms in patients with Type 2 diabetes.

DETAILED DESCRIPTION:
A high prevalence of gastrointestinal (GI) symptoms exist in both type 1 and type 2 diabetes that affect the quality of life negatively and substantially, although the underlying pathophysiology and relationship with glycemic control remain unclear. The current study aims to investigate if altering the microbiome though Pendulum T2D dietary supplementation can further enhance the efficacy of the current treatment while reducing the GI associated symptoms in patients with Type 2 diabetes mellitus who are already on a stable dose of metformin alone and/or alongside other oral or injectable anti-hyperglycemic agents (sulfonylurea agents, DPPIV inhibitor,Glucagon-like peptide (GLP)-1 agonist, sodium-glucose cotransporter (SGLT)-2 inhibitor and/or insulin) and with present GI symptoms. The study is a single site, prospective, open label, observational, single arm trial in 30 patients with type 2 diabetes with GI complaints using 1 or more oral or injectable anti-hyperglycemic agent and an HbA1C between 6.5% and 9.5%. The study will be 8 weeks in duration (2 weeks baseline and 6 weeks product intervention), with an option to continue to 6 months for those willing to continue taking the dietary supplement. As the study is observational and the data are to be used to for the purpose of evaluating improvement in GI symptoms during the intervention with Pendulum T2D there is no specific method to determine sample size.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index ≤ 45 kg/m2.
* Subjects with type 2 diabetes that are on a stable dose of one or more injectable or oral antihyperglycemia agents for at least 8 weeks prior to screening.
* HbA1c ≥ 6.5 % and ≤ 9.5% obtained at the screening visit.
* Subjects with any gastrointestinal symptoms including but not limited to heartburn, indigestion, diarrhea, constipation.
* Must be willing and be able to give written informed consent.

Exclusion Criteria:

* Type 1 diabetes
* Pregnant, nursing or planning pregnancy
* Planning elective surgery in the next 8 weeks
* Current or planned use of steroids, orally or injected
* Diagnosis of irritable bowel disease , diverticulitis, other significant GI illness
* Co-existing severe health condition, such as active cancer or unstable cardiovascular disease/congestive heart failure.
* Severe allergy to tape or any component of the CGM device

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-01-15 (Estimated); Primary Completion 2022-02-14 (Estimated); Study Completion 2022-06-14 (Estimated)

PRIMARY OUTCOMES:
Decreased Gastrointestinal Symptoms | 6 weeks
  Mean change from baseline in overall Gastrointestinal Symptom Rating Scale (GSRS) scores. The GSRS is a 15-item self-administered questionnaire related to abdominal pain, reflux, indigestion, diarrhea and constipation syndromes, that assesses the impact of gastrointestinal symptoms during the past week on a scale from 1 (no discomfort at all) to 7 (very severe discomfort).

SECONDARY OUTCOMES:
Increased time in glucose range | 6 weeks
  Measured by continuous glucose monitor (CGM)
Decreased time in hyperglycemic range | 6 weeks
  Measured by continuous glucose monitor (CGM)
Decreased time in hypoglycemic range | 6 weeks
  Measured by continuous glucose monitor (CGM)
Improvement in A1C | 6 weeks
  Point of Care Hemoglobin A1c (HbA1c) %
Improvement in fructosamine level | 6 weeks
  Blood draw to measure fructosamine
Improvement in A1C | 12 weeks
  Point of Care Hemoglobin A1c (HbA1c) %
Improvement in A1C | 24 weeks
  Point of Care Hemoglobin A1c (HbA1c) %

CONTACTS AND LOCATIONS:
Overall Officials: Anne L Peters, MD, Principal Investigator — University of Southern California
Locations (1):
- USC Westside Center for Diabetes, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No